CLINICAL TRIAL: NCT03864523
Title: Effect of Pioglitazone Administered to Patients With Adrenomyeloneuropathy: a Phase II, Single-arm, Multicentric Clinical Trial
Brief Title: Effect of Pioglitazone Administered to Patients With Adrenomyeloneuropathy
Acronym: XAMNPIOP2011
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pujol, Aurora, M.D. (Individual)
Collaborators: Instituto de Salud Carlos III (Other Government); Fundacion Hesperia (Other); ELA España Association (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XAMNPIOAP2011
Record Dates: First submitted 2016-09-16; First posted 2019-03-06 (Actual); Last update posted 2019-09-10 (Actual); Status verified 2019-03

CONDITIONS: Adrenomyeloneuropathy; X-linked Adrenoleukodystrophy
Keywords: AMN; pioglitazone
MeSH Terms: conditions — Adrenoleukodystrophy | interventions — Pioglitazone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- XAMNPIO (Experimental): Pioglitazone 15 mg tablets 2/day during 2 years
  Interventions: Drug: Pioglitazone

INTERVENTIONS:
Drug: Pioglitazone

SUMMARY:
X-linked adrenoleukodystrophy is a rare, demyelinating and neurodegenerative disorder, due to loss of function of a fatty acid transporter, the peroxisomal ABCD1 protein. Its more frequent phenotype, the adrenomyeloneuropathy in adults, is characterized by axonal degeneration in spinal cord, spastic paraparesis and a disabling peripheral neuropathy. Actually, there is no efficient treatment for the disease. The work of the researchers in the last twelve years dissecting the physiopathological basis of the disorder has uncovered an involvement of the early oxidative stress in the neurodegenerative cascade and mitocondrial depletion. In a preclinical trial they have observed that pioglitazone, a PPARγ/PGC-1α axis metabolic activator with immunomodulatory, anti-inflammatory and antioxidant response regulator properties, efficiently reverse the clinical symptoms and the axonal degeneration in the mouse model for the disease and normalize stress and mitochondrial depletion biomarkers.

The researchers will test the effectiveness of the drug in terms of motor function and correction of oxidative damage markers in proteins and DNA and inflammation markers in an open trial. Fifteen-twenty patients will be included and clinically explored and assessed in the HU of Bellvitge and the HU of Donostia using clinical scales for spasticity, evoked potentials, electroneurinograms and cranial RMN. The information will be collected in a data base that will be of great value to improve the present attention and the future follow-up of the patients and to facilitate their inclusion in therapeutic randomized, double blind, against placebo, multicentric and international clinical trials.

DETAILED DESCRIPTION:
Proof of concept for this trial is provided by the results of biochemical, neuropathological and motor effects of pioglitazone in two mouse models of AMN. Pioglitazone was given orally (9 mg/kg/day) for two months in both models.

The Abcd1-null mouse model already shows at 3,5 months biochemical signs oxidative stress that increase with time and are then associated with energy homeostasis alterations, although first clinical signs of AMN-i.e. axonopathy and locomotor impairment-appear at 20 months. In these mice, there are mitochondrial anomalies, decreased levels of PGC-1α which is a master regulator of mitochondrial biogenesis, and decreased levels and activity of SIRT1α, which activates PGC-1α.

The Abcd1-null mouse can be considered as a "AMN-like" model, because of the absence of demyelinating lesions in brain and spinal cord, the presence of non-inflammatory ''dying-back'' axonopathy in peripheral nerves and spinal cord and its late-onset motor deficits that all are hallmarks of AMN in X-ALD patients. This model was used to assess the efficacy of pioglitazone on several biochemical markers in the spinal cord of Abcd1-null mice (N=12), using comparisons with placebo-¬treated Abcd1-null mice (N=12) or wild-type mice (N=12).

In Abcd1-null mice treated with pioglitazone at 10,5 months of age and studied at 12 months (1,5 months following the beginning of the ongoing treatment), mitochondrial anomalies were corrected to the level of wild type control mice. Indeed, mitochondrial DNA and protein (including PGC-1α, NRF1 and TFAM) levels were corrected; as well as mitochondrial metabolism, as assessed by pyruvate kinase activity, ATP and NAD+ concentrations. Pioglitazone had no effect on SIRT1 expression (mRNA and protein levels). However, pioglitazone significantly lowered the carbonylation of SIRT1 protein, which presumably accounts for the observed rescue of SIRT1 activity.

In these mice treated with pioglitazone, oxidative lesions in the spinal cord were reversed. Studied oxidative stress biomarkers included markers of oxidative lesions to proteins (GSA, AASA), lipids (MDAL) and carbohydrates (CEL). Additionally, the activity and concentration level of antioxidant enzymes GPX1, which were increased in untreated Abcd1-null mice, but not SOD2, was normalized to the level of wild type mice.

The second mouse model is the double knockouts (DKO) in which both Abcd1 and Abcd2 transporters are inactivated. The Abcd1-/Abcd2-/-DKO exhibits greater VLCFA accumulation in spinal cord (Pujol et al., 2004), higher levels of oxidative damage to proteins, and a more severe AMN-¬like pathology, with earlier onset of motor impairment than the single Abcd1-null mouse (12 months in the DKO compared to 20 months in Abcd1-null mice). Efficacy of pioglitazone at the motor and neuropathologic levels was studied in 17 Abcd1-/Abcd2-/-mice comparing them with placebo-treated Abcd1-/Abcd2-/-mice (N=17) and wild-type mice (N=25).

In Abcd1-/Abcd2-/-mice treated with pioglitazone at 13 months of age and studied at 15 or 17 months (treatment duration of 2 to 4 months), axonal degeneration was prevented, as shown by the normalization to the control level of number of APP or synaptophysin positive axons.

Also, pioglitazone arrested the progression of locomotor deficits in these mice, as assessed by the treadmill test and the bar-cross test. Indeed, the locomotor performances of pioglitazone DKO after four months of treatment mice reached the performances of the controls.

Overall, these studies show the efficacy of treatment with pioglitazone in "AMN-like mice "and provide a strong rationale for conducting a preliminary open clinical trial with pioglitazone in AMN patients.

ELIGIBILITY:
Inclusion Criteria:

* Clinical signs of AMN with at least pyramidal signs in the lower limbs and difficulties to run.
* Presence of motor deficit according to the EDSS scale
* Ability to perform the 2MWT
* Normal brain MRI or brain MRI showing abnormalities that can be observed in AMN patients without cerebral form of X-ALD with a maximum Loes score of 4
* Ejection fraction > 50% at echocardiogram
* Normal electrocardiogram
* Normal urine cytology
* Normal liver function, as assessed by plasma ASAT, ALAT, PAL, γGT, bilirubin measures (≤2.5-fold normal values)
* Normal kidney function as assessed by plasma urea, creatinin (≤ 2-fold normal values)
* Appropriate steroid replacement if adrenal insufficiency is present
* Informed consent
* Affiliated to the Spanish Public Health System

Exclusion Criteria:

* Gadolinium enhancement on T1 sequence of any abnormal hypersignal of white matter, including myelinated pyramidal tracts, visible at brain MRI on FLAIR sequences
* Brain MRI abnormalities of the "AMN type" with a Loes score > 4
* Any abnormal hypersignal of white matter visible on FLAIR sequences other than of "AMN type" and related to X-ALD
* Patients taking pioglitazone or another glitazone during the past 6 months
* Diabetic patients (type I or II)
* Fasting blood glucose > 125 mg/L
* Glycosylated hemoglobin > 6%
* History of heart failure
* Heart failure (NYHA III to IV) or ejection fraction ≤ 50%
* History of cardiac disease
* [Hemoglobin] < 13g/dl in males, <12 g/dl in women
* Absolute neutrophil count (ANC) <1500 cells/mm3
* Platelet count <100,000 cells/mm3
* Significant peripheral edema (2+ or more on the Assessment Chart for Pitting Edema) of the extremities of any etiology
* Any evolutive malignancy during the last five years
* Prior or current bladder cancer
* Smokers (one pack/ day or more for at least 20 years), current or former
* Women with history of osteoporosis
* Menopaused woman with T-score < -2.5 on osteodensitometry measurement
* Any evolutive medical disease other than AMN
* Any psychiatric disease
* Pregnant or breastfeeding woman
* Either no pre-menopaused woman or no menopaused woman not taking any contraceptive method
* Hereditary intolerance to galatose, or malabsorption of glucose or galactose due the presence of monohydrated lactose.
* Hypersensibility to the active substance or to galactose (excipient)
* Concomitant treatment with cytochrome P450 CYP 2C8 inhibitors (e.g. gemfibrozil) or inducers (e.g. rifampicin)
* Taking of either vitamin A, E or lipoic acid during the past 3 months
* Contraindications for MRI procedure such as subjects with paramagnetic materials in the body, such as aneurysm clips, pacemakers, intraocular metal or cochlear implants
* Present participation to another therapeutic clinical trial for ALD
* Not easily contactable by the investigator in case of emergency or not capable to call the investigator
* Gross hematuria of unknown origin

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2016-01; Primary Completion 2019-03 (Actual); Study Completion 2019-07 (Actual)

PRIMARY OUTCOMES:
2 Minute Walk Test (2MWT) | 24 months
  The score at this test corresponds to the distance traveled by the patient during 2 minutes, on a flat surface

SECONDARY OUTCOMES:
Timed Up and Go (TUG) test | 24 months
  It consists in standing up, walking 3 meters, turning around, walk back to the chair and sitting back down, at regular pace
Time to walk 25 Feet (TW25) | 24 months
  In this test the patient should walk 7.62 meters (25 feet) as quickly, but safely, as possible without running
6 Minute Walk Test (6MWT) | 24 months
  It measures the distance an individual is able to walk over a total of six minutes on a hard, flat surface
Sensory disturbances: tactile | 24 months
  For the evaluation the Total Neuropathy Score (TNS) will be used (0-4)
Sensory disturbances: painful | 24 months
  For the evaluation the Total Neuropathy Score (TNS) will be used (0-4)
Sensory disturbances: vibratory | 24 months
  For the evaluation the Total Neuropathy Score (TNS) will be used (0-4)
Expanded disability status scale (EDSS) | 24 months
  This scale measures motor function, ranging from 0 (normal neurological examination) to 10 (death)
Dynamometer test (optional) | 24 months
  It measures the muscle strength
Ashworth scale | 24 months
  The Modified Ashworth Scale measures spasticity in patients who have lesions of the CNS or neurological disorders. The modified Ashworth scale ranges from 0 (no increase in tone) to 4 (Affected part(s) rigid in flexion or extension)
SF-Qualiveen | 24 months
  It measures the impact of urinary disorders in patients with neurological conditions
Revised Faecal Incontinence Scale (RFIS) | 24 months
  The RFIS is a short, reliable and valid five item scale used to asses faecal incontinence and to monitor patient outcomes following treatment. Response options are framed as 5-point Likert-type scales, with 0 indicating no impact of faecal incontinence problems on health-related quality of life and 4 indicating a high adverse impact. The RFIS total score is calculated by adding a person's score for each question. Adding the score for each of the five questions results in a possible score range of 0-20
Conventional MRI | 24 months
  FLAIR and T2 sequences may show subtle anomalies evaluated using the Loes scoring system. This MRI severity scale has been designed specifically for X-linked adrenoleukodystrophy and has been shown to correlate with severity of neurologic deficits and to be predictive of disease progression. Different brain regions are considered in the MRI severity score. Each area is scored as 0 if normal, 0.5 if unilateral involvement, and 1 if the lesion or atrophy is bilateral. The maximum severity score is 34; a score of 1 is considered abnormal.
Diffusion tensor Imaging (DTI) | 24 months
  Apparent diffusion coefficient (ADC) and fractional anisotropy (FA) will be measured
Brain MRI spectroscopy (MRS) | 24 months
  NAA/creatine and choline/creatine ratios will be measured
Nerve conduction studies: conduction velocity in the peroneal nerve | 24 months
  m/s
Nerve conduction studies: amplitude of the signal in the peroneal motor nerve | 24 months
  (mV)
Nerve conduction studies: conduction velocity in the sura sensitive nerve | 24 months
  (m/s)
Nerve conduction studies: amplitude of the signal in the sura sensitive nerve | 24 months
  (μV)
Motor Evoked Potentials (MEP): F wave | 24 months
  (ms) in right and left upper limb and right and left lower limb
Motor Evoked Potentials (MEP): Central latency | 24 months
  (ms) in right and left upper limb and right and left lower limb
Motor Evoked Potentials (MEP): Amplitude | 24 months
  (μV) in right and left upper limb and right and left lower limb
Motor Evoked Potentials (MEP): Central motor conduction time | 24 months
  (ms) in right and left upper limb and right and left lower limb
Somatosensory Evoked Potentials (SSEP): Latency N9 | 24 months
  (ms) right and left arms
Somatosensory Evoked Potentials (SSEP): Latency N13 | 24 months
  (ms) right and left arms
Somatosensory Evoked Potentials (SSEP): Latency N20 | 24 months
  (ms) right and left arms
Somatosensory Evoked Potentials (SSEP): Amplitude N20 | 24 months
  (μV) right and left arms
Somatosensory Evoked Potentials (SSEP): Latency N8 | 24 months
  (ms) right and left legs
Somatosensory Evoked Potentials (SSEP): Latency N22 | 24 months
  (ms) right and left legs
Somatosensory Evoked Potentials (SSEP): Latency P40 | 24 months
  (ms) right and left legs
Somatosensory Evoked Potentials (SSEP): Amplitude N40 | 24 months
  (μV) right and left legs
Brainstem Auditory Evoked Potentials (BAEP): Latency I wave | 24 months
  (ms) right and left
Brainstem Auditory Evoked Potentials (BAEP): Latency III wave | 24 months
  (ms) right and left
Brainstem Auditory Evoked Potentials (BAEP): Latency V wave | 24 months
  (ms) right and left
Brainstem Auditory Evoked Potentials (BAEP): Latency I-III wave | 24 months
  (ms) right and left
Brainstem Auditory Evoked Potentials (BAEP): Latency III-V wave | 24 months
  (ms) right and left
Brainstem Auditory Evoked Potentials (BAEP): Latency I-V wave | 24 months
  (ms) right and left
Markers of oxidative stress: GSA | 24 months
  Glutamic semialdehyde (GSA) will be measured in plasma. Results will be expressed in μmol/mol lysine
Markers of oxidative stress: CEL | 24 months
  Carboxyethyl-lysine (CEL) will be measured in plasma. Results will be expressed in μmol/mol lysine
Markers of oxidative stress: MDAL | 24 months
  N2-malondialdehyde-lysine (MDAL) will be measured in plasma. Results will be expressed in μmol/mol lysine
Markers of oxidative stress: CML | 24 months
  N2-carboxymethyl-lysine (CML) will be measured in plasma. Results will be expressed in μmol/mol lysine
Markers of oxidative stress: 8-oxoDG | 24 months
  7,8-dihydro-8-oxo-2-deoxyguanosine (8-oxoDG) will be measured in urine. Results will be expressed in ng/mg creatine
Markers of inflammation: HGF | 24 months
  HGF will be measured in plasma. Results will be expressed in pg/ml
Markers of inflammation: IL6 | 24 months
  IL6 will be measured in plasma. Results will be expressed in pg/ml
Markers of inflammation: IL8 | 24 months
  IL8 will be measured in plasma. Results will be expressed in pg/ml
Markers of inflammation: MCP-1 | 24 months
  MCP-1 will be measured in plasma. Results will be expressed in pg/ml
Markers of inflammation: NGF | 24 months
  NGF will be measured in plasma. Results will be expressed in pg/ml
Markers of inflammation: TNF | 24 months
  TNF will be measured in plasma. Results will be expressed in pg/ml
Markers of inflammation: adiponectin | 24 months
  Adiponectin will be measured in plasma. Results will be expressed in μg/ml
Markers of inflammation: CCR3 | 24 months
  CCR3 will be measured in RNA from peripheral mononuclear cells. Results will be expressed as relative gene expression
Markers of inflammation: CXCL5 | 24 months
  CXCL5 will be measured in RNA from peripheral mononuclear cells. Results will be expressed as relative gene expression
Markers of inflammation: CXCL9 | 24 months
  CXCL9 will be measured in RNA from peripheral mononuclear cells. Results will be expressed as relative gene expression
Markers of inflammation: IL9R | 24 months
  IL9R will be measured in RNA from peripheral mononuclear cells. Results will be expressed as relative gene expression
Markers of inflammation: PPARd | 24 months
  PPARd will be measured in RNA from peripheral mononuclear cells. Results will be expressed as relative gene expression
Markers of inflammation: GPX4 | 24 months
  GPX4 will be measured in RNA from peripheral mononuclear cells. Results will be expressed as relative gene expression
Markers of inflammation: STAT1 | 24 months
  STAT1 will be measured in RNA from peripheral mononuclear cells. Results will be expressed as relative gene expression

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - Bellvitge University Hospital, L'Hospitalet de Llobregat, Barcelona
  - Donostia University Hospital, Donostia / San Sebastian

IPD SHARING:
Plan to Share IPD: No